CLINICAL TRIAL: NCT00102661
Title: Continuous Infusion of Campath-1H Followed by Subcutaneous Injections in Previously Treated Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Berlex Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-424
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAMPATH-1H (Experimental): 15 mg infused daily for continuous infusion x 7 days; starting day 10, CAMPATH-1H 30 mg subcutaneously three times weekly for 11 additional weeks.
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H — 15 mg daily infused over 24 hours, continuous infusion x 7 days (Days 1 through 7). Each 15 mg dose prepared daily, immediately prior to starting the infusion. Starting day 10, CAMPATH-1H administered at dose of 30 mg subcutaneously three times weekly for 11 additional weeks.
  Other Names: Alemtuzumab; Campath

SUMMARY:
The goal of this clinical research study is to learn if giving CAMPATH-1H first as an injection into a vein, then as an injection under the skin can shrink or slow the growth of the disease in patients with chronic lymphocytic leukemia (CLL) who have already received standard therapy. Another goal is to learn if the side effects related to CAMPATH-1H treatment are less severe by giving the drug first as an injection into a vein then as an injection under the skin.

DETAILED DESCRIPTION:
The purposes of this trial are:

1. To evaluate the response rate (CR+PR) to CAMPATH-1H given as continuous infusion followed by subcutaneous injection in patients with previously treated CLL who have failed fludarabine therapy.
2. To evaluate whether CAMPATH-1H, given as a continuous infusion followed by subcutaneous injections to patients with previously treated CLL will improve tolerability of the agent and permit higher doses to be delivered through that route.
3. To evaluate the pharmacokinetics of CAMPATH-1H when given as a 24 hour continuous infusion followed by a subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years (CLL does not occur in the pediatric population).
* Signed informed consent.
* World Health Organization (WHO) performance status of 0, 1, or 2.
* Patients with B-CLL who have received fludarabine and are either refractory to frontline therapy or have relapsed within six months from receiving fludarabine-based therapy. Patients previously treated with Campath-1H are eligible.
* Serum creatinine <= 2mg/dL, total bilirubin <= 2mg/dL, and SGPT <= 3x upper limit of normal (ULN) unless due to direct infiltration of the liver or kidney with malignant cells.

Exclusion Criteria:

* Past history of anaphylaxis, following exposure to rat or mouse derived CDR-grafted humanized monoclonal antibodies.
* Prior chemotherapy, immunotherapy, or hormonal therapy within 2 weeks prior to study start. Hormonal replacement therapy is permitted. Prior therapy with monoclonal antibodies for at least 4 weeks prior to study start.
* Pregnant or nursing women or any patient of childbearing age unwilling to practice an acceptable form of contraception.
* Patients with history of HIV positivity.
* Active secondary malignancy.
* Active uncontrolled infection or any major systemic or other illness that would, in the opinion of the investigator, interfere with the patient's ability to comply with the protocol, compromise patient safety or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response Rate (CR+PR) to CAMPATH-1H | 3 months
  Rate is number of patients with CR+PR response to CAMPATH-1H where CR is Complete Response and PR is Partial Response RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org